CLINICAL TRIAL: NCT05481125
Title: Clareon Toric vs Eyhance Toric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILS241-P002
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cataract; Aphakia
Keywords: Cataracts; Phacoemulsification; IOL
MeSH Terms: conditions — Cataract; Aphakia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clareon/Clareon Toric (Experimental): Phacoemulsification surgery, followed by implantation with Alcon Clareon Aspheric Hydrophobic Acrylic IOL or Alcon Clareon Aspheric Hydrophobic Acrylic Toric IOL, as indicated. The second eye surgery is recommended to occur within 14 days after the 1st eye surgery.
  Interventions: Device: Clareon IOL; Device: Clareon Toric IOL; Procedure: Phacoemulsification surgery
- Eyhance/Eyhance Toric (Active Comparator): Phacoemulsification surgery, followed by implantation with TECNIS Eyhance IOL or TECNIS Eyhance Toric II IOL, as indicated. The second eye surgery is recommended to occur within 14 days after the 1st eye surgery.
  Interventions: Device: Eyhance IOL; Device: Eyhance Toric IOL; Procedure: Phacoemulsification surgery

INTERVENTIONS:
Device: Clareon IOL — Alcon Clareon Aspheric Hydrophobic Acrylic IOL for the visual correction of aphakia in adult patients in whom a cataractous lens has been removed. The lens is indicated for primary implantation in the capsular bag in the posterior chamber of the eye, replacing the natural crystalline lens. IOLs are implantable medical devices and are intended for long-term use over the lifetime of the pseudophakic subject.
  Other Names: Model SY60WF
  Arms: Clareon/Clareon Toric
Device: Clareon Toric IOL — Clareon Toric Aspheric Hydrophobic Acrylic Toric IOL for the visual correction of aphakia with pre-existing corneal astigmatism in adult patients in whom a cataractous lens has been removed. The lens is indicated for primary implantation in the capsular bag in the posterior chamber of the eye, replacing the natural crystalline lens. IOLs are implantable medical devices and are intended for long-term use over the lifetime of the pseudophakic subject.
  Other Names: Models CNW0T3, CNW0T4, CNW0T5, CNW0T6 as available
  Arms: Clareon/Clareon Toric
Device: Eyhance IOL — TECNIS Eyhance IOL with TECNIS Simplicity Delivery System for the visual correction of aphakia in adult patients in whom a cataractous lens has been removed by extracapsular cataract extraction. The lens is intended to be placed in the capsular bag. IOLs are implantable medical devices and are intended for long-term use over the lifetime of the pseudophakic subject.
  Other Names: Model DIB00
  Arms: Eyhance/Eyhance Toric
Device: Eyhance Toric IOL — TECNIS Eyhance Toric II IOL with TECNIS Simplicity Delivery System for the visual correction of aphakia and pre-existing corneal astigmatism of one diopter or greater in adult patients with or without presbyopia in whom a cataractous lens has been removed by phacoemulsification and who desire reduction in residual refractive cylinder. The lens is intended to be placed in the capsular bag. IOLs are implantable medical devices and are intended for long-term use over the lifetime of the pseudophakic subject.
  Other Names: Models DIU150, DIU225, DIU300, DIU375 as available
  Arms: Eyhance/Eyhance Toric
Procedure: Phacoemulsification surgery — Cataract removal by routine small incision phacoemulsification surgery

SUMMARY:
The primary purpose of this study is to compare the Clareon/Clareon Toric Intraocular Lenses (IOLs) to the Eyhance/Eyhance Toric IOLs in binocular Best Corrected Distance Visual Acuity (BCDVA) at 3 months postoperative.

DETAILED DESCRIPTION:
This study will enroll adults 22 years of age and older diagnosed with cataracts in both eyes with planned bilateral cataract removal by routine small incision phacoemulsification surgery. Subjects will attend up to 7 scheduled visits: A screening visit, two operative visits, and four post-operative visits. The expected individual duration of participation in the study is 3 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Planned bilateral cataract removal by routine small incision phacoemulsification surgery;
* Planned implantation of either test or comparator IOL (per randomization) in at least one eye with approximately 1.00 - 3.00 diopter (D) of preoperative corneal astigmatism;
* Predicted postoperative astigmatism of ≤ 0.5 D in both operative eyes based on a Toric calculator;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any disease or pathology, other than cataract, that (in the investigator's opinion) may reduce potential Best Corrected Distance Visual Acuity (BCDVA) to a level worse than 0.2 logarithm minimum angle of resolution (logMAR);
* Clinically significant (in the investigator's opinion) corneal pathology, dry-eye or ocular surface disease that would adversely affect a) the biometry measures and/or toric calculations and b) the visual outcome;
* History of previous intraocular or corneal surgery (including laser-assisted in situ keratomileusis (LASIK));
* Any other planned ocular surgical procedures including but not limited to limbal relaxing incision (LRI), astigmatic keratotomy, LASIK, and retinal laser treatment within the study time frame;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Seeta Eye Centers, Poughkeepsie, New York
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina
  - Vision for Life, Nashville, Tennessee
  - Houston Eye Associates, Houston, Texas
  - Berkeley Eye Center, Houston, Texas
  - Texas Eye Research Center, Hurst, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 investigative sites located in the United States.
Pre-assignment Details: Of the 203 enrolled, 14 subjects were exited prior to randomization as screen failures, and 14 subjects were discontinued after randomization and prior to attempted implantation. This reporting group includes all subjects with attempted implantation per actual treatment (175).
Groups:
- Clareon/Clareon Toric: Phacoemulsification surgery, followed by implantation with Alcon Clareon Aspheric Hydrophobic Acrylic IOL or Alcon Clareon Aspheric Hydrophobic Acrylic Toric IOL, as indicated. The second eye surgery was recommended to occur within 14 days after the 1st eye surgery.
- Eyhance/Eyhance Toric: Phacoemulsification surgery, followed by implantation with TECNIS Eyhance IOL or TECNIS Eyhance Toric II IOL, as indicated. The second eye surgery was recommended to occur within 14 days after the 1st eye surgery.
Period: Overall Study
Arm/Group | Clareon/Clareon Toric | Eyhance/Eyhance Toric
Started (Randomized with attempted implantation) | 89 | 86
First Eye Implanted | 89 | 86
Second Eye Implanted | 86 | 84
Completed | 88 | 84
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Implanted Analysis Set (AAS): All eyes with successful study IOL implantation and with at least one postoperative visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clareon/Clareon Toric | Eyhance/Eyhance Toric | Total
Number analyzed (Participants) | 89 | 86 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (7.63) | 70.4 (7.73) | 69.7 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 54 | 101
  Male | 42 | 32 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 77 | 74 | 151
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 70 | 74 | 144
  Black or African American | 15 | 9 | 24
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 89 | 86 | 175

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Best-corrected Distance Visual Acuity (BCDVA) at 4 Meters Under Bright Lighting Conditions
Description: Visual acuity was tested at a distance of 4 meters using a refraction chart and the correction obtained from a manifest refraction. BCDVA was measured in logarithm minimum angle of resolution (logMAR) units, with 0.00 logMar equating to 20/20 Snellen, which is considered normal distance eyesight. A lower logMAR value (more negative value) indicates better eyesight. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Month 3 postoperative visit
Population: AAS with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon/Clareon Toric | Eyhance/Eyhance Toric
Number analyzed (Participants) | 86 | 81
logMAR | -0.100 (0.0880) | -0.055 (0.0716)
Statistical Analysis 1: Comparison: Clareon/Clareon Toric vs Eyhance/Eyhance Toric; Test type: Non-Inferiority — Non-inferiority margin = 0.1 logMAR; Since a non-inferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the non-inferiority margin; Mean Difference (Final Values) = -0.045, 95% CI 1-sided [upper limit -0.024], Standard Error of Mean 0.0125 — Mean difference (Clareon/Clareon Toric minus Eyhance/Eyhance Toric). Upper Confidence Limit is presented

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent until study exit. The total expected duration of participation for each subject was approximately 3 months.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is included with unit of "eyes." The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting group. This analysis population includes all eyes with attempted IOL implantation (successful or aborted after contact with the eye) as treated.
Groups:
- Pretreatment: All subjects in the safety analysis set prior to initiation of treatment
- Clareon/Clareon Toric First Eye: All first study eyes implanted with Clareon/Clareon Toric IOL
- Clareon/Clareon Toric Second Eye: All second study eyes implanted with Clareon/Clareon Toric IOL
- Clareon/Clareon Toric Systemic: All subjects implanted with Clareon/Clareon Toric IOL
- Eyhance/Eyhance Toric First Eye: All first study eyes implanted with Eyhance/Eyhance Toric IOL
- Eyhance/Eyhance Toric Second Eye: All second study eyes implanted with Eyhance/Eyhance Toric IOL
- Eyhance/Eyhance Toric Systemic: All subjects implanted with Eyhance/Eyhance Toric IOL
Arm/Group | Pretreatment | Clareon/Clareon Toric First Eye | Clareon/Clareon Toric Second Eye | Clareon/Clareon Toric Systemic | Eyhance/Eyhance Toric First Eye | Eyhance/Eyhance Toric Second Eye | Eyhance/Eyhance Toric Systemic
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/89 | 0/86 | 0/89 | 0/86 | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/175 | 2/89 | 0/86 | 2/89 | 2/86 | 0/84 | 3/86
Other Adverse Events (participants affected / at risk) | 0/175 | 11/89 | 8/86 | 0/89 | 6/86 | 7/84 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=175) | Clareon/Clareon Toric First Eye (N=89) | Clareon/Clareon Toric Second Eye (N=86) | Clareon/Clareon Toric Systemic (N=89) | Eyhance/Eyhance Toric First Eye (N=86) | Eyhance/Eyhance Toric Second Eye (N=84) | Eyhance/Eyhance Toric Systemic (N=86)
Ciliary zonular weakness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iris disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular lens repositioning (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=175) | Clareon/Clareon Toric First Eye (N=89) | Clareon/Clareon Toric Second Eye (N=86) | Clareon/Clareon Toric Systemic (N=89) | Eyhance/Eyhance Toric First Eye (N=86) | Eyhance/Eyhance Toric Second Eye (N=84) | Eyhance/Eyhance Toric Systemic (N=86)
Posterior capsule opacification (Eye disorders) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 6 (6) | 5 (5) | 0 (0) | 5 (5) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT05481125/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT05481125/SAP_001.pdf